CLINICAL TRIAL: NCT03610087
Title: Technology-Enabled Collaborative Care for Youth (TECC-Y): A Feasibility Study
Brief Title: Technology-Enabled Collaborative Care for Youth
Acronym: TECC-Y
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Medical Psychiatry Alliance (Other); Trillium Health Centre (Other); The Hospital for Sick Children (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Peter Selby, Deputy Physician-in-Chief- Education|Clinician Scientist|Chief, Medicine in Psychiatry Division|CAMH|, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 121-2017
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Psychosis; Metabolic Disease; Cardiovascular Risk Factor
MeSH Terms: conditions — Psychotic Disorders; Metabolic Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Intensity Intervention (Other): The comparison group (low intensity) receives access to the e-platform and given an educational package with information about nutrition, physical activity, and smoking based on the NAVIGATE program (Mueser et al., 2015); i.e., a comprehensive program for implementing coordinated speciality care) with weekly e-mail reminders for 12 weeks. Participants receive access to online resources and free online webinars about these healthy behaviours.
  Interventions: Behavioral: Low Intensity Intervention
- High Intensity Intervention (Experimental): The intervention group (high intensity) receives a technology-enabled CCM intervention. Participants receive access to an online platform and infographic modules to learn more about nutrition, physical activity, and smoking cessation. Also, they are assigned a personal health coach who collaboratively schedules weekly virtual sessions via the platform to discuss the educational materials, goal setting and motivation, and provide support in the 12-week program. The participant's health coach reviews the participant's concerns and goals weekly with a virtual care team (VCT; including a psychiatrist, addictions specialist, nutrition specialist, peer mentor, and recreational therapist), who provides individualized recommendations to include in the participant's treatment plan. Participants have access to online resources and online webinars about nutrition, physical activity and smoking.
  Interventions: Behavioral: High Intensity Intervention

INTERVENTIONS:
Behavioral: Low Intensity Intervention — Participants will have access via the online platform to the NAVIGATE self-help modules for physical activity, nutrition and quitting smoking with a list of community resources. Subjects will be sent a standard reminder emails once per week to complete their modules and connect with their main provider for any assistance.
  Arms: Low Intensity Intervention
Behavioral: High Intensity Intervention — Participants will receive individualized treatment planning, in collaboration with a Care Coordinator, and the Virtual Care Team (VCT). Interactive modules on physical activity, nutrition and quitting smoking will be provided via the online platform. the virtual team will be engaged to provide treatment and/or recommendations regarding the following: increasing physical activity, improving nutrition and diet, smoking cessation (psychosocial support plus medications), and medication adherence. Participants in this arm will have weekly check-ins with their assigned Care Coordinator where they will be able to discuss VCT recommendations, and progress on their goals.
  Other Names: TECC-Y
  Arms: High Intensity Intervention

SUMMARY:
The overall objective is to develop scalable interventions to address the physical health needs of patients affected by early psychosis. The objective of this project is to conduct a feasibility study of a high intensity technology-enabled collaborative care model (CCM) compared to lower intensity self-help modules and email support for early identification and treatment of cardio-metabolic risk factors in youth, ages 16-29, affected by early psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Ages 16 - 29 years
* Clinician diagnosis of early psychosis (diagnosed in last 5 years)
* Prescribed psychiatric medication, stable for 4 weeks
* Access to telephone or internet through computer or mobile

Exclusion Criteria:

* Unable to provide consent
* Unable to understand English

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in patient engagement | Baseline, 6-weeks, 12-weeks, and 24-weeks.
  The primary outcome is patient engagement will be defined as participant activation in the program measured via self-report levels of perceived benefit from the program.

SECONDARY OUTCOMES:
Healthy Behaviour Change | Baseline, 6-weeks, 12-weeks, and 24-weeks.
  The secondary outcome is to explore whether a CCM will help facilitate healthy behavioral changes in physical activity, nutrition, and smoking.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Selby P, Vojtila L, Ashfaq I, Dragonetti R, Melamed OC, Carriere R, LaChance L, Kohut SA, Hahn M, Mulsant BH. Technology-enabled collaborative care for youth with early psychosis: A protocol for a feasibility study to improve physical health behaviours. Early Interv Psychiatry. 2021 Aug;15(4):828-836. doi: 10.1111/eip.13018. Epub 2020 Aug 3. PMID 32748501